CLINICAL TRIAL: NCT05483842
Title: Effects of Reiki on Heart Rhythm, Biochemistry, Cortisol Findings and Anxiety in Individuals With Arrhythmia: A Randomized Prospective, Single-Blind and Placebo-Controlled Study
Brief Title: Reiki Effects on Heart Rhythm, Biochemistry and Cortisol Findings, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E.60364
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Heart Diseases
Keywords: Reiki; Heart Rhythm; Arrythmia; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Heart Diseases; Arrhythmias, Cardiac | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients did not know which group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki Group (Experimental): Personal Information Form (PIF) and Beck Anxiety Scale (BAS) were administered to the Reiki group through face-to-face interviews. Then, blood was taken for biochemical blood and cortisol findings and ECG was taken. After the pre-tests of the patients were completed, the application was made under the guidance of a researcher with a Usui Reiki Master & Teacher degree and by a researcher with Reiki II training. In accordance with the Reiki Practice Protocol, an empty and silent room was selected in the hospital. Reiki was applied one-on-one to energy centers (crown chakra, forehead chakra, throat chakra, heart chakra, solar plexus, sacral region, root chakra, knees, ankle and feet) for 30 minutes. On the second day, 30 minutes of distant Reiki was applied. BAS was administered 1 week later; ECG was taken and biochemistry blood was taken.
  Interventions: Other: Reiki
- Sham Reiki Group (Placebo Comparator): Personal Information Form (PIF) and Beck Anxiety Scale (Scale) were administered to this group by face-to-face interviews. Then, blood was taken for biochemical blood and cortisol findings and ECG was taken. After the pre-tests of the patients were completed. The Sham Reiki group was practiced by a student nurse who did not receive Reiki training by imitating the hand positions used in Reiki practice. Before the applications, the researcher, the student was told about aura equalization and chakras, the student only imitated gestures and facial expressions, but did not give Reiki energy to the patients. BAS was administered 1 week later; ECG was taken and biochemistry blood was taken.
  Interventions: Other: Sham Reiki
- Control Group (No Intervention): Personal Information Form (PIF) and Beck Anxiety Scale (BAS) were administered to this group by face-to-face interviews. Then, blood was taken for biochemical blood and cortisol findings and ECG was taken. After 1 week, BAS, blood tests and ECG have applied again.

INTERVENTIONS:
Other: Reiki — Consisting of the words "rei" meaning "spirit" and "ki" meaning "universal life force", Reiki means spiritually directed life force energy. Reiki practice has an important place in modern medicine and the nursing profession because it cures many diseases resistant to known treatments, has no side effects, is easy to apply, is safe, effective and economical.
  In the Reiki method, which is one of the complementary and alternative methods, energy is transferred through the hands. Its basis is based on the principle that when there is a blockage in an energy center, disease occurs and the energy transferred by touching, strengthens and heals the body's self-healing ability by opening the blockages. Reiki practitioners who have received training and initiation perform the practice by holding their hands in certain positions on the recipient's body.
  Arms: Reiki Group
Other: Sham Reiki — Sham means to pretend; therefore, in this study, the sham Reiki placebo provider pretended to perform a Reiki session by moving her hands on the patient's body in a specific order for a 30-minute period following strictly operationalized measures.
  Arms: Sham Reiki Group

SUMMARY:
This study aimed to investigate the effects of Reiki, which is a complementary and traditional method, on heart rhythm, biochemistry and cortisol findings, and anxiety in individuals with arrhythmia.

DETAILED DESCRIPTION:
Reiki has an essential place in modern medicine and the nursing profession because it cures many diseases resistant to known treatments, has no side effects, is easy to apply, and is safe, effective, and economical. In the Reiki method, the energy is transferred through the hands, and a care provider nurse is a tool that performs their profession by touching in patient care and also shares the universal life energy, transferring the flowing and formed energy. When the literature is reviewed, there are a limited number of studies in which Reiki affects heart rate, cortisol level, and vital signs. However, there are not enough studies examining the effects of heart patients' symptoms, anxiety, and their condition on Reiki results. In this context, this study aimed to investigate the effects of Reiki energy on heart rhythm, biochemistry, cortisol findings, and anxiety in people with arrhythmia.

The study was conducted as a pretest-posttest, randomized prospective, single-blind and placebo-controlled. The study was conducted with patients who applied to a training and research hospital with arrhythmia complaints between April 5 and June 30, 2022. The data was collected using "Personal Information Form (PIF)" and "Beck Anxiety Scale (BAS)". Also, biochemical tests and cortisol findings and ECG (Electrocardiography) analyses were assessed.

PIF and BAS were applied to patients who agreed to participate in the study and met the inclusion criteria. Then blood was drawn for biochemical tests and cortisol findings and EKG was taken. Patients were randomized 1:1 into groups by a single therapist at a single institution according to a parallel design. There were three treatment arms in the study: Reiki treatment (n=22), Sham Reiki treatment (placebo)(n=22), and a control group with no treatment (n=22). A second-degree Reiki practitioner applied Reiki to the energy centers for 30 minutes in the Reiki group. On the second day, distant Reiki was also conducted for 30 minutes. The Sham Reiki group, on the other hand, was handled similarly to the Reiki practice by a student who had not been trained in Reiki. In the control group, nothing was done. One week later, BAS was applied to all patients, blood was drawn for biochemical testing and an ECG was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* No communication problem
* Diagnosed with cardiac arrhythmia
* Who agree to participate in the Reiki practice
* Who is competent to answer the data collection tools to be used in the research
* Patients who have not used complementary practices in the last six months

Exclusion Criteria:

* Reiki practitioner or trainer,
* Have received energy therapies such as Reiki/therapeutic touch,
* Patients who were diagnosed with another disease during the research process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Change from Sodium values at a week | -Within 1 hour of first admission. -A week later.
  In this section, there is Sodium value required for the normal electrical activity of the heart.
Change from Potassium values at a week | -Within 1 hour of first admission. -A week later.
  In this section, there is Potassium value required for the normal electrical activity of the heart.
Change from Calcium values at a week | -Within 1 hour of first admission. -A week later.
  In this section, there is Calcium value required for the normal electrical activity of the heart.
Change from Magnesium values at a week | -Within 1 hour of first admission. -A week later.
  In this section, there is Magnesium value required for the normal electrical activity of the heart.
Change from Baseline Cortisol at a week | -Within 1 hour of first admission. -A week later.
  In addition, individuals with arrhythmia experience stress and have a blood cortisol value due to the relationship between stress and cortisol hormone.
Change from Baseline Heart Rhythm at a week | -Within 1 hour of first admission. -A week later.
  In order to determine cardiac arrhythmias, 12-lead ECG was taken from the individuals within the scope of the study.
Change from Baseline Beck Anxiety Scale at a week | -Within 1 hour of first admission. -A week later.
  The scale measured the frequency of anxiety symptoms and signs experienced by the individual. The scale is a Likert-type scale consisting of 21 items and scores between 0-3. The minimum score to be taken from the scale is 0 and the maximum score is 63. As the score obtained from the scale increases, the anxiety of the individual increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay BEKTAS AKPINAR, PhD, Principal Investigator — Ankara Medipol University
Locations (1):
- Nursemin Ünal, Ankara, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Gallob R. Reiki: a supportive therapy in nursing practice and self-care for nurses. J N Y State Nurses Assoc. 2003 Spring-Summer;34(1):9-13. PMID 14639776
- [Background] Rao A, Hickman LD, Sibbritt D, Newton PJ, Phillips JL. Is energy healing an effective non-pharmacological therapy for improving symptom management of chronic illnesses? A systematic review. Complement Ther Clin Pract. 2016 Nov;25:26-41. doi: 10.1016/j.ctcp.2016.07.003. Epub 2016 Aug 2. PMID 27863608
- [Background] Thrane S, Cohen SM. Effect of Reiki therapy on pain and anxiety in adults: an in-depth literature review of randomized trials with effect size calculations. Pain Manag Nurs. 2014 Dec;15(4):897-908. doi: 10.1016/j.pmn.2013.07.008. Epub 2014 Feb 28. PMID 24582620
- [Background] McManus DE. Reiki Is Better Than Placebo and Has Broad Potential as a Complementary Health Therapy. J Evid Based Complementary Altern Med. 2017 Oct;22(4):1051-1057. doi: 10.1177/2156587217728644. Epub 2017 Sep 5. PMID 28874060
- [Background] Morero JAP, Pereira SS, Esteves RB, Cardoso L. Effects of Reiki on Mental Health Care: A Systematic Review. Holist Nurs Pract. 2021 Jul-Aug 01;35(4):191-198. doi: 10.1097/HNP.0000000000000456. PMID 34115737
- [Background] Bat N. The effects of reiki on heart rate, blood pressure, body temperature, and stress levels: A pilot randomized, double-blinded, and placebo-controlled study. Complement Ther Clin Pract. 2021 May;43:101328. doi: 10.1016/j.ctcp.2021.101328. Epub 2021 Feb 17. PMID 33639516
- [Derived] Bektas Akpinar N, Ozcan Yuce U, Cansiz G, Yurtsever D, Ozkanat C, Unal N, Sabanoglu C, Altinbas Akkas O, Yurtsever S. Is Reiki effective in reducing heart rhythm, cortisol levels, and anxiety and improving biochemical parameters in individuals with cardiac disease? Randomized placebo-controlled trial. Eur J Cardiovasc Nurs. 2024 Oct 21;23(7):771-779. doi: 10.1093/eurjcn/zvae051. PMID 38652801